CLINICAL TRIAL: NCT00841893
Title: Effects of a Specific Spice on Energy Expenditure, Substrate Oxidation, Appetite and Energy Intake
Brief Title: Effects of a Specific Spice on Energy Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Nikolaj Ture Gregersen/Ph.D.student, Department of Human Nutrition, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: B253-IHE-spice2-NTG
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: Thermogenesis; Meal-induced thermogenesis; Energy expenditure; Fat oxidation; Carbohydrate oxidation; Bioactive ingredient; Spice
MeSH Terms: interventions — Amines

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Mustard
  Interventions: Dietary Supplement: Mustard (dijon)
- 2 (Experimental): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mustard (dijon) — The specific spice added to a brunch meal
  Arms: 1
Dietary Supplement: Placebo — Placebo added to a brunch meal
  Arms: 2

SUMMARY:
The objective of this study is to examine whether a specific spice is capable of affecting energy metabolism.

Since chili and other spices have been shown to increase energy expenditure and in some cases also affect energy intake/appetite compared to placebo, the investigators expect that the specific spice may actually increase energy expenditure and potentially also decrease appetite - although not to a large degree.

DETAILED DESCRIPTION:
Several pungent food ingredients, such as chili, and also other bioactive food ingredients, e.g. green tea, have been shown to be able to increase energy expenditure and fat oxidation during the hours following a meal containing the bioactive ingredient. Furthermore, we will also look at the subjects own feelings of appetite and thereby examine whether the appetite is affected by the spicy food, since a few studies have suggested an effect of bioactive ingredients on appetite/energy intake. We expect to see some small effects on these parameters.

ELIGIBILITY:
Inclusion Criteria:

* male
* healthy and not using medication (regularly)
* normal weight
* non-smoker
* tolerate and like spicy food
* stable body weight last two months

Exclusion Criteria:

* increased blood pressure
* mental, metabolic and chronic diseases

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Energy expenditure (resting)/Meal-induced thermogenesis | November 2008

SECONDARY OUTCOMES:
VAS-scores for different appetite parameters (incl. satiety, hunger, fullness, prospective food intake, well-being, thirst etc.) | November 2008
Blood pressure | November 2008
Heart rate | November 2008
Substrate oxidation (fat and carbohydrate) | November 2008

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Professor MD, Study Chair — Department of Human Nutrition, Faculty of Life Sciences, University of Copenhagen
Locations (1):
- Department of Human Nutrition, Faculty of Life Sciences, university of Copenhagen, Frederiksberg C, Copenhagen, Denmark